CLINICAL TRIAL: NCT04822870
Title: Comparison of Ultrasound-guided Quadratus Lumborum Block and Iliohypogastric/Ilioinguinal Nerve Block for Postoperative Pain Management in Patients Undergoing Cesarean Section: a Randomized Double-blind Clinical Trial Study
Brief Title: Comparison of Ultrasound-guided Quadratus Lumborum Block and Iliohypogastric/Ilioinguinal Nerve Block for Postoperative Pain Management in Patients Undergoing Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, Head of Anesthesiology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-Z-01
Record Dates: First submitted 2021-03-17; First posted 2021-03-30 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Quadratus Lumborum Block; Iliohypogastric/Ilioinguinal Nerve Block; Cesarean Section
MeSH Terms: interventions — Analgesia, Epidural

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- quadratus lumborum block (Experimental): Parturients receive ultrasound-guided quadratus lumborum block as post-operative analgesia.
  Interventions: Procedure: quadratus lumborum block
- iliohypogastric/ilioinguinal nerve block (Experimental): Parturients receive ultrasound-guided iliohypogastric/ilioinguinal nerve block as post-operative analgesia.
  Interventions: Procedure: iliohypogastric/ilioinguinal nerve block
- epidural analgesia (Active Comparator): Parturients receive epidural morphine via epidural catheter placed during anesthesia as post-operative analgesia.
  Interventions: Procedure: epidural analgesia

INTERVENTIONS:
Procedure: quadratus lumborum block — Quadratus lumborum block is an effective nerve block method in post-cesarean section analgesia. It is a relatively new technique that may provide analgesic effect in somatic pain and visceral pain, but has not been verified yet.
  Arms: quadratus lumborum block
Procedure: iliohypogastric/ilioinguinal nerve block — Iliohypogastric/ilioinguinal nerve block is a widely used nerve block technique. It can provide somatic analgesia effect in post-cesarean section.
  Arms: iliohypogastric/ilioinguinal nerve block
Procedure: epidural analgesia — Epidural analgesia is a traditional analgesia method. Epidural morphine can provide effective analgesia but may cause plenty adverse effect.
  Arms: epidural analgesia

SUMMARY:
The purpose of this study is to compare the analgesic effect of ultrasound-guided quadratus lumborum block and iliohypogastric/ilioinguinal nerve block for postoperative pain management in patients undergoing cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* gestation of at least 37 weeks
* American Society of Anesthesiologists (ASA) physical status I or II
* finish Pfannenstiel section under combined spinal and epidural anesthesia

Exclusion Criteria:

* pruritus existed before the surgery
* allergic to lidocaine, ropivacaine or dexamethasone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
morphine consumption | 24 hours postoperatively
  Every parturient use a patient-controlled intravenous analgesia pump as supplement for the interventions. The analgesia pump contains morphine and can record morphine consumption. Postoperative use of morphine can reflect analgesic effect.

SECONDARY OUTCOMES:
morphine consumption | 6 hours postoperatively
  Every parturient use a patient-controlled intravenous analgesia pump as supplement for the interventions. The analgesia pump contains morphine and can record morphine consumption. Postoperative use of morphine can reflect analgesic effect.
morphine consumption | 12 hours postoperatively
  Every parturient use a patient-controlled intravenous analgesia pump as supplement for the interventions. The analgesia pump contains morphine and can record morphine consumption. Postoperative use of morphine can reflect analgesic effect.
morphine consumption | 48 hours postoperatively
  Every parturient use a patient-controlled intravenous analgesia pump as supplement for the interventions. The analgesia pump contains morphine and can record morphine consumption. Postoperative use of morphine can reflect analgesic effect.
pain score | 6 hours postoperatively
  Use visual analogue scale (VAS) 0-10 to evaluate pain intensity and reflect analgesic effect. 0 refers to completely no pain, 10 refers to the most severe pain she has experienced.
pain score | 12 hours postoperatively
  Use visual analogue scale (VAS) 0-10 to evaluate pain intensity and reflect analgesic effect. 0 refers to completely no pain, 10 refers to the most severe pain she has experienced.
pain score | 24 hours postoperatively
  Use visual analogue scale (VAS) 0-10 to evaluate pain intensity and reflect analgesic effect. 0 refers to completely no pain, 10 refers to the most severe pain she has experienced.
pain score | 48 hours postoperatively
  Use visual analogue scale (VAS) 0-10 to evaluate pain intensity and reflect analgesic effect. 0 refers to completely no pain, 10 refers to the most severe pain she has experienced.
effective analgesia time | 48 hours postoperatively
  Time period between finish the intervention and the first time parturient use the patient-controlled intravenous analgesia pump for analgesia supplement.
adverse effect | 6 hours postoperatively
  Nausea and vomiting, pruritus, oversedation, respiratory depression and urinary retention are considered adverse effects. The incidence and severity are recorded, 1 score refers to mild, 2 scores refers to moderate, 3 scores refers to severe and treatment needed.
adverse effect | 12 hours postoperatively
  Nausea and vomiting, pruritus, oversedation, respiratory depression and urinary retention are considered adverse effects. The incidence and severity are recorded, 1 score refers to mild, 2 scores refers to moderate, 3 scores refers to severe and treatment needed.
adverse effect | 24 hours postoperatively
  Nausea and vomiting, pruritus, oversedation, respiratory depression and urinary retention are considered adverse effects. The incidence and severity are recorded, 1 score refers to mild, 2 scores refers to moderate, 3 scores refers to severe and treatment needed.
adverse effect | 48 hours postoperatively
  Nausea and vomiting, pruritus, oversedation, respiratory depression and urinary retention are considered adverse effects. The incidence and severity are recorded, 1 score refers to mild, 2 scores refers to moderate, 3 scores refers to severe and treatment needed.
satisfaction score | 48 hours postoperatively
  Ask the patient to evaluate satisfaction score using 0-10. 0 refers totally dissatisfied, 10 refers to the most satisfied
hospital stay | at discharge assessed up to 10 days
  The hospitalize length
hospitalize cost | at discharge assessed up to 10 days
  Total cost in this hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Yi Feng, MD, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China